CLINICAL TRIAL: NCT01527019
Title: A Phase III Non-Inferiority Open-label Multicenter Randomized Clinical Trial to Compare CEPHALOSPORIN to NORFLOXACIN in the Treatment of Acute Cystitis
Brief Title: Comparison in the Treatment of Acute Cystitis Using Cephalosporin and Norfloxacin (CECI)
Acronym: CECI
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: the company suspended the persecution of this combination
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF125
Record Dates: First submitted 2012-01-31; First posted 2012-02-06 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2012-02

CONDITIONS: Cystitis
Keywords: Acute Cystitis
MeSH Terms: conditions — Cystitis | interventions — Norfloxacin; Cephalosporins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cephalosporin oral suspension (Experimental): 130 research subjects on cephalosporin oral suspension (test) 400 mg once daily
  Interventions: Drug: Cephalosporins
- Cephalosporin capsules (Experimental): 130 research subjects on cephalosporin capsules (test) 400 mg once daily
  Interventions: Drug: Cephalosporins
- Norfloxacin (Active Comparator): 130 research subjects on norfloxacin (test) 400 mg twice daily
  Interventions: Drug: Norfloxacin

INTERVENTIONS:
Drug: Norfloxacin — Norfloxacin Pills, 400 mg twice daily. Treatment time will range according to sex and age (male and elderly subjects will receive 7 days of treatment, while female subjects who are 18-59 years old will receive 3 days of treatment)
  Arms: Norfloxacin
Drug: Cephalosporins — Cephalosporins Caps, 400 mg once daily. Treatment time will range according to sex and age (male and elderly subjects will receive 7 days of treatment, while female subjects who are 18-59 years old will receive 3 days of treatment)
  Arms: Cephalosporin capsules
Drug: Cephalosporins — Cephalosporins Oral Suspension, 400 mg once daily. Treatment time will range according to sex and age (male and elderly subjects will receive 7 days of treatment, while female subjects who are 18-59 years old will receive 3 days of treatment)
  Arms: Cephalosporin oral suspension

SUMMARY:
This study is to assess if the efficacy of cephalosporin is similar to the efficacy of norfloxacin in the acute cystitis treatment.

ELIGIBILITY:
Inclusion Criteria:

* Sign, initialize and date the informed consent form
* Age ≥ 18 years
* For urinary infection diagnosis, the following parameters must be considered in the urine I test:
* Leukocyturia: ≥ 15,000 leukocytes
* Epidermal cells: < 20,000/mL
* Presence of bacteriuria
* Presence of nitrite (positive results)
* To have a 2 points score (from 12 points) regarding the following symptoms of acute cystitis:
* Dysuria
* Urinary urgency
* Frequent urination
* Pain in the upper area of pubis

Each symptom must be scored according to the classification below. Total score may range from 0 to 12 points.

Severity Value Absent 0 Mild 1 Moderate 2 Severe 3

Exclusion Criteria:

Research subjects that meet any of the criteria below will not be eligible for the study:

* Asymptomatic urinary infection or infection in any organ
* Documented incidence of UTI in the last year
* Symptoms of pyelonephritis (cystitis symptoms plus fever, lower back pain or chills)
* History of complicated urinary tract infection (congenital abnormalities, urinary tract distortion or obstruction, formation of calculus in the urinary tract)
* Use of catheter in the urinary tract
* Chronic renal or hepatic disease
* Seizure-related diseases
* Neurological deficits that interfere in the urinary flow and tract defense
* Decompensated diabetes mellitus (fasting blood glucose ≥ 150 mg/dL);
* Immunodepression:
* Subjects with the human immunodeficiency virus (HIV)
* Chronic use of corticosteroids in a dose ≥ 5 mg/day of prednisone for over 30 days
* Any diseases related to immune dysfunction
* Severe comorbidities (at the investigator's discretion)
* History of allergy to penicillins, cephalosporines or quinolones
* Subjects on medications such as antibiotics, amiodarone, antacids or sucralphate, tricyclic antidepressants, antipsychotics, cyclosporine, cisapride, didanosine, erythromycin, fembufeno, gliburide (a sulphonilurea), nitrofurantoin, probenecid, procainamide, quinidine, sotalol, teophylline, warfarin
* Treatment due to UTI two weeks before entering study, or on antimicrobial treatment at least 3 times within the last 12 months
* Use of phenazopyridine 7 days before entering the study
* Hospitalization 30 days before study enrollment
* Female research subjects that are pregnant, breastfeeding, or women with childbearing potential that deny to use at least two safe contraceptive methods during study
* Participation in another clinical trial in the last 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-10; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Bacteriological Eradication | 5-9 days
  The primary endpoint of this study will be the bacteriological eradication rate obtained 5-9 days following the end of the treatment with study drugs.

SECONDARY OUTCOMES:
Clinical Cure | bacteriological eradication rate 4-6 weeks; clinical cure rate 5-9 days; clinical cure rate 4-6 weeks;uroculture 5-9 days and 4-6 weeks
  To determine the bacteriological eradication rate 4-6 weeks after the end of treatment; To determine the clinical cure rate 5-9 days after the end of treatment; To determine the clinical cure rate 4-6 weeks after the end of treatment; To determine the clinical cure rate for research subjects with negative uroculture 5-9 days and 4-6 weeks after the end of treatment; To assess the research subjects adherence to the study treatment; To assess the safety of antibiotics according to the incidence of adverse events and serious adverse events.